CLINICAL TRIAL: NCT04058990
Title: A 2:1 Randomized Trial Comparing the Agent Paclitaxel-Coated PTCA Balloon Catheter vs SeQuent Please Drug Eluting Balloon Catheter for the Treatment of a Small Vessel De Novo Native Coronary Artery Lesion.
Brief Title: Safety and Effectiveness of Agent Paclitaxel-Coated PTCA Balloon Catheter. (AGENT Japan SV)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S2313
Record Dates: First submitted 2019-08-08; First posted 2019-08-16 (Actual); Results first posted 2022-12-23 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Masking Description: SV study: A prospective, multicenter, 2:1 randomized, controlled, single-blind, non-inferiority trial.150 subjects are expected to be enrolled to support a 2:1 randomization. (Investigational test device: Agent DCB, N=100 subjects or Control device: SeQuent Please DCB, N=50 subjects)
  ISR substudy: A prospective, multicenter, single-arm, open-label trial. 30 subjects are expected to be enrolled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Agent Paclitaxel-Coated PTCA Balloon Catheter (Experimental): Treatment of a Small Vessel De Novo Native Coronary Artery Lesion with a paclitaxel-coated balloon. (Agent Paclitaxel-Coated PTCA Balloon Catheter with paclitaxel 2.0 μg/mm²)
  Interventions: Device: Device: Paclitaxel-Coated PTCA Balloon Catheter
- SeQuent Please Drug Eluting Balloon Catheter (Active Comparator): Treatment of a Small Vessel De Novo Native Coronary Artery Lesion with a paclitaxel-coated balloon. (SeQuent Please Drug Eluting Balloon Catheter with paclitaxel 3.0 μg/mm²)
  Interventions: Device: SeQuent Please Drug Eluting Balloon Catheter with Paclitaxel

INTERVENTIONS:
Device: Device: Paclitaxel-Coated PTCA Balloon Catheter — Percutaneous Transluminal Coronary Angioplasty
  Arms: Agent Paclitaxel-Coated PTCA Balloon Catheter
Device: SeQuent Please Drug Eluting Balloon Catheter with Paclitaxel — Percutaneous Transluminal Coronary Angioplasty
  Arms: SeQuent Please Drug Eluting Balloon Catheter

SUMMARY:
A Randomized Trial Comparing the Agent Paclitaxel-Coated PTCA Balloon Catheter vs SeQuent Please Drug Eluting Balloon Catheter for the Treatment of a Small Vessel De Novo Native Coronary Artery Lesion.

DETAILED DESCRIPTION:
Primary objective is to evaluate the safety and effectiveness of the Agent ™ Paclitaxel-Coated PTCA Balloon Catheter for the treatment of Japanese subjects with a small vessel de novo native atherosclerotic coronary artery lesion or in-stent restenosis (ISR) of a previously treated lesion.

Primary endpoint: Target Lesion Failure (TLF) rate at 6 months post index-procedure. TLF is defined as any ischemia driven revascularization of the target lesion (TLR), myocardial infarction (MI, Q-wave and non-Q-wave) related to the target vessel, or cardiac death.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be at least 20 years of age.
2. Subject understands the trial requirements and the treatment procedures and provides written informed consent before any study-specific tests or procedures are performed.
3. Subject is eligible for percutaneous coronary intervention (PCI).
4. Subject has documented stable angina pectoris or unstable angina pectoris. If subject has documented stable angina pectoris, one of the following criteria meet.

   * ≥90% diameter stenosis.
   * Stenosis that is considered a cause of stable effort angina (Only when it's without confirmation of significant stenosis).
   * Stenosis that is confirmed a cause of functional ischemia with any test.
5. Subject is an acceptable candidate for coronary artery bypass grafting (CABG).
6. Subject is willing to comply with all protocol-required follow-up evaluation.
7. Patients undergoing first or second treatment for ISR lesions for the non-randomized ISR substudy.
8. The target lesion meets all following criteria.

   * Target lesion length must measure (by visual estimate) ≤28 mm.
   * Target lesion must be a visually estimated reference vessel diameter (RVD) ≥2.00mm and <3.00 mm (This applys for SV trial. For ISR substudy: RVD ≥2.00mm and ≤4.00 mm.).
   * Target lesion must be a de novo lesion located in a native coronary artery with visually estimated stenosis ≥75% and <100% (This applys for SV trial. For ISR substudy: Target lesion for ISR must be in-stent restenosis of a previously-treated lesion located in a native coronary artery with visually estimated stenosis ≥75% and <100%.).
   * Coronary anatomy is likely to allow delivery of an investigational device to the lesions.
   * Target lesion must be successfully pre-dilated.
9. Planned treatment of 2 coronary artery lesions in 2 vessels may be treated (For SV trial, up to two lesions per vessel can be treated. For ISR substudy, single lesion per vessel can be treated.).

Exclusion Criteria:

1. Subject has had an acute myocardial infarction within 72 hours prior to the index procedure.
2. Subject has cardiogenic shock, hemodynamic instability requiring inotropic or mechanical circulatory support, intractable ventricular arrhythmia, or ongoing intractable angina.
3. Subject has severe left ventricular dysfunction with ejection fraction <30%.
4. Subject has received an organ transplant or is on a waiting list for an organ transplant.
5. Subject is receiving or scheduled to receive chemotherapy within 30 days before or after the index procedure.
6. Subject has renal failure with a serum creatinine of > 2.0mg/dL or who is receiving dialysis or chronic immunosuppressant therapy.
7. Subjects has one of the following.

   * Not expected to live for the duration of the study (1 year) by investigator's discretion due to other serious medical illness.
   * Current problems with substance abuse.
   * Planned procedure that may cause non-compliance with the protocol or confound data interpretation.
8. Planned PCI (including staged procedures) or CABG after the index procedure.
9. Subject previously treated at any time with intravascular brachytherapy.
10. Subject has a known allergy to contrast and/or the investigational device or protocol-required concomitant medications, iopromide, raw materials of Agent DCB and SeQuent Please DCB, P2Y12 inhibitor or aspirin).
11. Subject has a platelet count <100,000 cells/mm3 or >700,000 cells/mm3.
12. Subject has a white blood cell (WBC) count < 3,000 cells/mm3.
13. Subject has documented or suspected liver disease, including laboratory evidence of hepatitis.
14. Subject has a history of bleeding diathesis or coagulopathy or will refuse blood transfusions.
15. Subject has had a history of cerebrovascular accident (CVA) or transient ischemic attack (TIA) within the past 6 months.
16. Subject has an active peptic ulcer or active gastrointestinal (GI) bleeding.
17. Target vessel has been treated with Paclitaxel Eluting Stent or Balloon prior to the index procedure.
18. Target vessel has been treated with any type of PCI within 6 months prior to the index procedure.
19. Target vessel requires the use of adjunctive primary treatment modalities immediately prior to investigational device's treatment.
20. Non-target vessel has been treated with any type of PCI within 24 hours prior to the index procedure.
21. Subject is participating in another investigational drug or device clinical trial that has not reached its primary endpoint.
22. Subject intends to participate in another investigational drug or device clinical trial within 6 months after the index procedure.
23. Subject with known intention to procreate within 6 months after the index procedure.
24. Subject is a woman who is pregnant or nursing.
25. Target lesion meets any of the following criteria:

    * Left main location.
    * Located within 5 mm of the origin of the left anterior descending (LAD) coronary artery or left circumflex (LCX) coronary artery by visual estimate.
    * > 50% stenosis of an additional lesion proximal or distal to the target lesion (by visual estimate).
    * Located within a saphenous vein graft or an arterial graft.
    * Will be accessed via a saphenous vein graft or an arterial graft.
    * Involves a complex bifurcation (e.g., bifurcations requiring treatment with more than 1 stent).
    * TIMI flow 0 (total occlusion) prior to wire crossing.
    * Excessive tortuosity proximal to or within the lesion.
    * Extreme angulation proximal to or within the lesion.
    * Target lesion and/or target vessel proximal to the lesion is severely calcified by visual estimate to expect sub-optimal balloon expansion.
    * Target lesion and/or target vessel adjacent to the target lesion presents with dissection or aneurysm by visual estimate.
    * Restenosis from previous intervention (This is applicable only to SV trial.).
    * PCI within 10 mm proximal or distal to the target lesion (by visual estimate) at any time prior to the index procedure （This is applicable only to SV trial.）.
    * Planned treatment of a single lesion with more than 1 investigational device.
    * In-stent restenosis due to stent fracture or recoil (This is applicable only to ISR substudy.).
26. Non-target lesion to be treated during the index procedure meets any of the following criteria:

    * Located in the target vessel (This is applicable only to ISR substudy.).
    * Located within a bypass graft (venous or arterial).
    * Left main location.
    * Chronic total occlusion.
    * Involves a complex bifurcation.
    * Located within 15 mm of the proximal or distal shoulder of the target lesion by visual estimate in the case of the same vessel with a target lesion for SV trial.
27. Subject has unprotected left main coronary artery disease (>50% diameter stenosis).
28. Thrombus, or possible thrombus, present in the target vessel.
29. Subject with known coronary artery spasm.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2019-12-12 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2026-06-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Masato Nakamura, MD, Principal Investigator — Toho University Ohashi Medical Center
Locations (14):
- Japan (14):
  - Kokura Memorial Hospital, Kitakyushu, Fukuoka
  - Sapporo Higashi Tokushukai Hospital, Sapporo, Hokkaido
  - Japan Labour Health and Welfare Organization Kanto Rosai Hospital, Kawasaki, Kanagawa
  - Shonan Kamakura General Hospital, Ōfuna, Kanagawa
  - Saiseikai Yokohama-City Eastern Hospital, Yokohama, Kanagawa
  - Kyoto-Katsura Hospital, Kyoto, Kyoto
  - Sendai Kousei Hospital, Sendai, Miyagi
  - Miyazaki Medical Association Hospital, Miyazaki, Miyazaki
  - Osaka Saiseikai Nakatsu Hospital, Kita, Osaka
  - Sakurabashi Watanabe Advanced Healthcare Hospital, Osaka, Osaka
  - Toho University Ohashi Medical Center, Meguro City, Tokyo
  - Showa Medical University Hospital, Shinagawa-Ku, Tokyo
  - Tokyo Women's Medical University Hospital, Shinjuku-Ku, Tokyo
  - Teikyo University Hospital, tabashi City, Tokyo

IPD SHARING:
Plan to Share IPD: No
The confidentiality of records/data obtained in the trial will remain anonymous for analysis and publication.
  The information and data, obtained from the trial is used without personal identification.

RESULTS

PARTICIPANT FLOW:
Groups:
- Agent Paclitaxel-Coated PTCA Balloon Catheter - Randomized; Agent DCB - Single Arm ISR Sub Study: Treatment of a Small Vessel De Novo Native Coronary Artery Lesion with a paclitaxel-coated balloon. (Agent Paclitaxel-Coated PTCA Balloon Catheter with paclitaxel 2.0 μg/mm²)
  Device: Paclitaxel-Coated PTCA Balloon Catheter: Percutaneous Transluminal Coronary Angioplasty
- SeQuent Please Drug Eluting Balloon Catheter - Randomized: Treatment of a Small Vessel De Novo Native Coronary Artery Lesion with a paclitaxel-coated balloon. (SeQuent Please Drug Eluting Balloon Catheter with paclitaxel 3.0 μg/mm²)
  SeQuent Please Drug Eluting Balloon Catheter with Paclitaxel: Percutaneous Transluminal Coronary Angioplasty
Period: Overall Study
Arm/Group | Agent Paclitaxel-Coated PTCA Balloon Catheter - Randomized | SeQuent Please Drug Eluting Balloon Catheter - Randomized | Agent DCB - Single Arm ISR Sub Study
Started | 101 | 49 | 30
Completed | 100 | 49 | 30
Not Completed | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Data are reported separately for each cohort as pooled mean and standard deviations across cohorts do not provide meaningful data.
Groups:
- Total: Total of all reporting groups
Arm/Group | Agent Paclitaxel-Coated PTCA Balloon Catheter - Randomized | SeQuent Please Drug Eluting Balloon Catheter - Randomized | Agent DCB - Single Arm ISR Sub Study | Total
Number analyzed (Participants) | 101 | 49 | 30 | 180
Age, Continuous [Mean (Standard Deviation); unit: years] — Data are reported separately for each cohort as pooled mean and standard deviations across cohorts do not provide meaningful data
  years
    Agent Paclitaxel-Coated PTCA Balloon Catheter - Randomized | 68.37 (10.62) | 0 (0) | 0 (0) | 68.37 (10.62)
    SeQuent Please Drug Eluting Balloon Catheter - Randomized | 0 (0) | 67.73 (10.38) | 0 (0) | 67.73 (10.38)
    Agent DCB - Single Arm ISR Sub Study | 0 (0) | 0 (0) | 68.50 (11.71) | 68.50 (11.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 38 | 26 | 139
  Male | 26 | 11 | 4 | 41
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 101 | 49 | 30 | 180
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 101 | 49 | 30 | 180
Stable Angina [Count of Participants; unit: Participants] | 98 | 45 | 29 | 172
Unstable Angina [Count of Participants; unit: Participants] | 3 | 4 | 1 | 8

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Events Included in the Primary Endpoint (Target Lesion Failure)
Description: TLF is defined as any ischemia driven revascularization of the target lesion (TLR), myocardial infarction (MI, Q-wave and non-Q-wave) related to the target vessel, or cardiac death.
Time Frame: 6 months post procedure
Population: Non-inferiority analysis - ITT population - all subjects who sign an Informed Consent Form, are enrolled in the trial, and are implanted with the assigned, randomized study device.
Measure: Count of Participants; unit: Participants
Arm/Group | Agent Paclitaxel-Coated PTCA Balloon Catheter | SeQuent Please Drug Eluting Balloon Catheter
Number analyzed (Participants) | 101 | 49
Participants | 3 | 0
Statistical Analysis 1: Comparison: Agent Paclitaxel-Coated PTCA Balloon Catheter vs SeQuent Please Drug Eluting Balloon Catheter; [Not Specified]; Test type: Non-Inferiority — 13.2% non-inferiority margin; p = 0.0012, Farrington-Manning

2. Other Pre Specified Outcome: Percentage of Participants With Events Included in the Primary Endpoint (Target Lesion Failure)
Description: as for outcome 1
Time Frame: 6 months post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Agent DCB - Single Arm ISR Sub Study
Number analyzed (Participants) | 30
Participants | 1

ADVERSE EVENTS:
Time Frame: 6 months following procedure
Arm/Group | Agent Paclitaxel-Coated PTCA Balloon Catheter | SeQuent Please Drug Eluting Balloon Catheter | Agent DCB - Single Arm ISR Sub Study
All-Cause Mortality (participants affected / at risk) | 0/101 | 0/49 | 1/30
Serious Adverse Events (participants affected / at risk) | 15/101 | 4/49 | 3/30
Other Adverse Events (participants affected / at risk) | 46/101 | 20/49 | 12/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Agent Paclitaxel-Coated PTCA Balloon Catheter (N=101) | SeQuent Please Drug Eluting Balloon Catheter (N=49) | Agent DCB - Single Arm ISR Sub Study (N=30)
Cardiac disorders (Cardiac disorders) | 7 (9) | 3 (3) | 2 (2)
Gastrointestinal disorders (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Hepatobiliary disorders (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Eye disorders (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Nervous system disorders (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Renal and urinary disorders (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Vascular disorders (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Agent Paclitaxel-Coated PTCA Balloon Catheter (N=101) | SeQuent Please Drug Eluting Balloon Catheter (N=49) | Agent DCB - Single Arm ISR Sub Study (N=30)
Cardiac disorders (Cardiac disorders) | 10 (13) | 5 (5) | 3 (3)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 13 (13) | 2 (2) | 0 (0)
General disorders and administration site conditions (Gastrointestinal disorders) | 8 (10) | 3 (4) | 3 (3)
Gastrointestinal disorders (General disorders) | 6 (8) | 3 (3) | 1 (2)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 7 (7) | 4 (4) | 2 (2)
Infections and infestations (Infections and infestations) | 7 (7) | 2 (2) | 2 (2)
Eye disorders (Eye disorders) | 3 (4) | 0 (0) | 1 (1)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 4 (4) | 0 (0) | 2 (2)
Vascular disorders (Vascular disorders) | 3 (3) | 4 (5) | 0 (0)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 3 (4)
Nervous system disorders (Nervous system disorders) | 3 (3) | 2 (2) | 1 (1)
Investigations (Investigations) | 2 (3) | 1 (1) | 3 (4)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1)
Ear and labyrinth disorders (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0)
Hepatobiliary disorders (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Psychiatric disorders (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Renal and urinary disorders (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Immune system disorders (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
[Not Specified]

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The restriction depends on the conditions on the Clinical Study Agreement at each site. The PI must notify the sponsor about the publication and receive the approval from the sponsor prior to any results/data relavant to the AGENT Japan trial to be in public.

DOCUMENTS (2):
  • Study Protocol (2020-09-30): https://cdn.clinicaltrials.gov/large-docs/90/NCT04058990/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-24): https://cdn.clinicaltrials.gov/large-docs/90/NCT04058990/SAP_001.pdf